CLINICAL TRIAL: NCT02121457
Title: Effects of Brazil Nuts Consumption on Selenium Status and Cognitive Performance in Older Adults With Mild Cognitive Impairment: a Randomized Controlled Pilot Trial
Brief Title: Brazil Nuts Effects on Selenium Status and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Barbara Rita Cardoso, Bárbara Rita Cardoso, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doutorado-2014
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Mild Cognitive Impairment
Keywords: cognitive performance; selenium; brazil nuts; oxidative stress
MeSH Terms: conditions — Cognitive Dysfunction | interventions — 2S albumin, brazil nut; Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): This group did not receive any intervention.
- Treatment Group (Experimental): This group took one Brazil nut daily during 6 months.
  Interventions: Dietary Supplement: Brazil nut; Dietary Supplement: selenium

INTERVENTIONS:
Dietary Supplement: Brazil nut — Participants of the treatment group were instructed to take one Brazil nut daily during 6 months. Brazil nuts were supplied in 2-month allowances at no cost together with written nutritional information and a calendar to monitor the compliance. Compliance was monitored in intervals of 2 months by checking the calendar and counting returned nuts. Compliance was considered to be adequate if ≥85% of Brazil nuts were consumed. All subjects were instructed to maintain their normal diet and to avoid additional Brazil nuts during the study.
  Arms: Treatment Group
Dietary Supplement: selenium
  Arms: Treatment Group

SUMMARY:
Some studies reported that selenium status is associated with cognitive function. However only a few reports have investigated whether selenium supplementation can benefit cognitive performance and in most of them selenium supplementation was not exclusive. Also, none of those reports have used foods rich in selenium as a source of supplementation. Thus, the aim of our study was to investigate whether the consumption of Brazil nuts improves cognitive function. We hypothesized that the daily consumption of Brazil nuts would have benefits on selenium status, increase antioxidant enzyme activity and improve cognitive function in older adults with MCI.

DETAILED DESCRIPTION:
We enrolled older patients with MCI who attended the Memory and Aging Unit of the Geriatrics Division, University of São Paulo Medical School (Brazil). All participants fulfilled the criteria proposed by the International Working Group on Mild Cognitive Impairment (Winblad et al., 2004), which include the following: (1) the person is neither normal nor demented; (2) there is evidence of cognitive deterioration shown by subjective report in conjunction with objective cognitive deficits; and (3) activities of daily living are preserved and complex instrumental functions are either intact or minimally impaired. The diagnosis of MCI was based on a comprehensive neuropsychological assessment which included the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) neuropsychological battery (Welsh et al., 1994; Bertolucci et al., 2001). Participants were recruited from May 2011 to August 2012. Eligible subjects were aged 60 years or older, fluent in Portuguese, and free of any other significant neurologic or psychiatric diseases. None of them presented major depression or psychosis, had a regular intake of Brazil nuts, used supplements with selenium, or had intolerance to oleaginous food. An informed consent was obtained before the interview from all participants. The research protocol was approved by the Research Ethics Comittee of the Faculdade de Ciências Farmacêuticas da Universidade de São Paulo.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or older,
* fluent in Portuguese,
* free of any other significant neurologic or psychiatric diseases

Exclusion Criteria:

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Selenium level in plasma and erythrocyte | 6 months

SECONDARY OUTCOMES:
cognitive performance | 6 months
  Cognitive performance was measured by using six sub-testes from the CERAD neuropsychological battery have been administered to assess fundamental cognitive abilities.

OTHER OUTCOMES:
Oxidative stress parameters | 6 months
  Oxidative stress was evaluated by measuring glutathione peroxidase activity, Oxygen radical absorbance capacity (ORAC) and Malondialdehyde (MDA).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia F Cozzolino, PhD, Study Director — University of Sao Paulo
Locations (1):
- University Of são Paulo, São Paulo, São Paulo, Brazil